CLINICAL TRIAL: NCT00308750
Title: A Randomized, Open-label Phase II Study of Pemetrexed (Alimta) Plus Carboplatin With or Without Enzastaurin Hydrochloride, or Docetaxel Plus Carboplatin as First Line Treatment in Patients With Advanced Stage Non-small Cell Lung Cancer (NSCLC)
Brief Title: First Line Chemotherapy Treatment of Advanced Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10651; H6Q-US-S004 (Other: Eli Lilly and Company)
Record Dates: First submitted 2006-03-28; First posted 2006-03-30 (Estimated); Results first posted 2021-05-13 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-04

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — enzastaurin; Pemetrexed; Docetaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Enzastaurin/Pemetrexed/Carboplatin (Experimental)
  Interventions: Drug: enzastaurin; Drug: pemetrexed; Drug: carboplatin
- Pemetrexed/Carboplatin (Experimental)
  Interventions: Drug: pemetrexed; Drug: carboplatin
- Docetaxel/Carboplatin (Active Comparator)
  Interventions: Drug: docetaxel; Drug: carboplatin

INTERVENTIONS:
Drug: enzastaurin — 1125-1200 milligrams (mg) loading dose then 500 mg, oral, daily, until disease progression
  Other Names: LY317615
  Arms: Enzastaurin/Pemetrexed/Carboplatin
Drug: pemetrexed — 500 milligrams per square meter (mg/m^2), intravenous (IV), once every (q) 21 days, six 21 day cycles or progressive disease
  Other Names: LY231514; Alimta
  Arms: Enzastaurin/Pemetrexed/Carboplatin; Pemetrexed/Carboplatin
Drug: docetaxel — 75 mg/m^2, IV, q 21 days, six 21 day cycles or progressive disease
  Arms: Docetaxel/Carboplatin
Drug: carboplatin — Area under the curve (AUC) 6, IV, q 21 days, six 21 day cycles or progressive disease

SUMMARY:
The purposes of this study are to determine:

The safety of enzastaurin plus pemetrexed with carboplatin, pemetrexed with carboplatin, or docetaxel with carboplatin and any side effects that might be associated with the combination of these drugs.

Whether the combination of enzastaurin plus pemetrexed and carboplatin or pemetrexed and carboplatin can help participants with non-small cell lung cancer (NSCLC) live longer, compared with the combination of docetaxel and carboplatin.

Whether the combination of enzastaurin plus pemetrexed and carboplatin or pemetrexed and carboplatin can make your tumor smaller or disappear, and for how long, compared with the combination of docetaxel and carboplatin.

The effects of enzastaurin plus pemetrexed with carboplatin, pemetrexed with carboplatin or docetaxel with carboplatin have on your disease related symptoms.

The relation of smoking history and hormone replacement therapy (for women only) may have to your lung cancer treatment results.

The effects of certain genes and proteins in samples of your blood and tumor tissue in order to learn more about NSCLC and how enzastaurin works in the body.

ELIGIBILITY:
Inclusion Criteria:

* You must have been diagnosed with NSCLC.
* You must be able to visit the doctor's office weekly during the active treatment period and as needed during the study follow-up period.
* You must be willing and able to swallow capsules.
* Your entry labs and medical tests must meet study requirements.
* You must be willing to have blood samples drawn and tissue samples obtained for gene and protein testing.

Exclusion Criteria:

* You have received radiation within 2 weeks of study enrollment.
* You have previously received any anti-cancer drug therapy for NSCLC.
* You have an active infection or other serious condition.
* You take aspirin or aspirin-like medication regularly and are not able to stop taking them for a few days during each cycle of chemotherapy.
* You have recently lost a significant amount of weight.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2006-03; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (4):
- United States (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Burlington, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chapel Hill, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Columbia, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Houston, Texas

REFERENCES:
- [Derived] Socinski MA, Raju RN, Stinchcombe T, Kocs DM, Couch LS, Barrera D, Rousey SR, Choksi JK, Jotte R, Patt DA, Periman PO, Schlossberg HR, Weissman CH, Wang Y, Asmar L, Pritchard S, Bromund J, Peng G, Treat J, Obasaju CK. Randomized, phase II trial of pemetrexed and carboplatin with or without enzastaurin versus docetaxel and carboplatin as first-line treatment of patients with stage IIIB/IV non-small cell lung cancer. J Thorac Oncol. 2010 Dec;5(12):1963-9. doi: 10.1097/JTO.0b013e3181fd42eb. PMID 21102260

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Presented in the participant flow are the reasons participants discontinued from study treatment.
Groups:
- Enzastaurin/Pemetrexed/Carboplatin: Enzastaurin loading dose of 1125 milligrams (mg) or 1200 mg orally on Day -7 (pre-chemotherapy) followed by 500 mg administered orally once daily starting from Day -6 until disease progression.
  Pemetrexed 500 milligrams per square meter (mg/m^2) and carboplatin [area under the curve (AUC)] 6 milligrams*minutes per milliliter (mg*min/mL) as an intravenous infusion on Day 1 every 21 days for a maximum of 6 cycles (21-day cycle) or disease progression whichever came first.
- Pemetrexed/Carboplatin: Pemetrexed 500 mg/m^2 and carboplatin AUC 6 mg*min/mL as an intravenous infusion on Day 1 every 21 days for a maximum of 6 cycles (21-day cycle) or disease progression whichever came first.
- Docetaxel/Carboplatin: Docetaxel 75 mg/m^2 and carboplatin AUC 6 mg*min/mL as an intravenous infusion on Day 1 every 21 days for a maximum of 6 cycles (21-day cycle) or disease progression whichever came first.
Period: Overall Study
Arm/Group | Enzastaurin/Pemetrexed/Carboplatin | Pemetrexed/Carboplatin | Docetaxel/Carboplatin
Started | 72 | 74 | 72
Received at Least 1 Dose of Study Drug | 67 | 72 | 70
Completed | 0 | 34 | 23
Not Completed | 72 | 40 | 49
Not completed — Adverse Event | 9 | 9 | 13
Not completed — Withdrawal by Subject | 6 | 2 | 3
Not completed — Physician Decision | 3 | 4 | 3
Not completed — Sponsor Decision | 1 | 0 | 0
Not completed — Disease Progression | 47 | 24 | 28
Not completed — Unrelated Complication | 3 | 0 | 1
Not completed — Death | 1 | 0 | 1
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — New Primary Disease Identified | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Enzastaurin/Pemetrexed/Carboplatin: Enzastaurin loading dose of 1125 mg or 1200 mg orally on Day -7 (pre-chemotherapy) followed by 500 mg administered orally once daily starting from Day -6 until disease progression.
  Pemetrexed 500 mg/m^2 and carboplatin AUC 6 mg*min/mL as an intravenous infusion on Day 1 every 21 days for a maximum of 6 cycles (21-day cycle) or disease progression whichever came first.
- Total: Total of all reporting groups
Arm/Group | Enzastaurin/Pemetrexed/Carboplatin | Pemetrexed/Carboplatin | Docetaxel/Carboplatin | Total
Number analyzed (Participants) | 72 | 74 | 72 | 218
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.2 (9.8) | 64.0 (10.0) | 64.0 (9.1) | 64.4 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 33 | 30 | 94
  Male | 41 | 41 | 42 | 124
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African | 5 | 11 | 8 | 24
  Caucasian | 62 | 63 | 63 | 188
  Hispanic | 5 | 0 | 1 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 72 | 74 | 72 | 218
Disease Stage at Study Entry [Count of Participants; unit: Participants] — Disease stage describes how big the tumor is and how far it has spread from the site of origin. Stages range from Stage I to Stage IV. Stage III is further separated into Stage IIIA and IIIB. Stage IIIB (cancer spread to distant lymph nodes and invaded other organs like heart, esophagus etc). Stage IV (cancer spread throughout the body).
  Participants
    Stage IIIB | 6 | 5 | 6 | 17
    Stage IV | 66 | 69 | 66 | 201

OUTCOME MEASURES:

1. Primary Outcome: Time to Disease Progression
Description: Time to disease progression was defined as the time from randomization to the first date of documented disease progression or death if the participant dies due to disease progression. Response was defined using Response Evaluation Criteria In Solid Tumors (RECIST, version 1.0) criteria. Progressive disease (PD) was defined as having at least a 20% increase in sum of the longest diameter of target lesions. For participants who have not had documented disease progression, time to disease progression was censored at the date of death or date of last visit. For participants who received other anti-tumor therapy prior to disease progression, time to disease progression was censored at the first available date of other anti-tumor therapy.
Time Frame: Baseline to measured PD up to 22.3 months
Population: All randomized participants. Twenty (20) participants in Enzastaurin/Pemetrexed/Carboplatin group, 15 participants in Pemetrexed/Carboplatin group, and 17 participants in Docetaxel/Carboplatin group were censored for analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enzastaurin/Pemetrexed/Carboplatin | Pemetrexed/Carboplatin | Docetaxel/Carboplatin
Number analyzed (Participants) | 52 | 59 | 55
months | 4.6 [3.2 to 6.7] | 6.0 [4.6 to 6.5] | 4.1 [2.6 to 6.3]
Statistical Analysis 1: Comparison: Enzastaurin/Pemetrexed/Carboplatin vs Docetaxel/Carboplatin; Test type: Superiority or Other; p = 0.40, Log Rank
Statistical Analysis 2: Comparison: Pemetrexed/Carboplatin vs Docetaxel/Carboplatin; Test type: Superiority or Other; p = 0.19, Log Rank

2. Secondary Outcome: Tumor Biomarkers Associated With Clinical Outcomes
Description: As specified in the protocol, tumor biomarker samples were collected from participants on the pemetrexed arms only but were not intended to be analyzed at the individual study level.
Time Frame: Baseline, Cycle 1, Cycle 2 (21-day cycle each), and 30-day post study treatment follow-up
Population: Zero participants were analyzed due to insufficient samples being collected.
Arm/Group | Enzastaurin/Pemetrexed/Carboplatin | Pemetrexed/Carboplatin | Docetaxel/Carboplatin
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Assessment of Smoking History (All Participants) and Hormone Replacement Therapy (Female Participants Only) Associated With Clinical Outcomes
Description: Data for smoking history and hormone replacement therapy were collected but were not intended to be analyzed at the individual study level.
Time Frame: Baseline
Population: Zero participants were analyzed due to insufficient samples being collected.
Arm/Group | Enzastaurin/Pemetrexed/Carboplatin | Pemetrexed/Carboplatin | Docetaxel/Carboplatin
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Number of Participants With Adverse Events (AEs) or Deaths
Description: Data presented are the number of participants who experienced 1 or more AEs or any serious AEs (SAEs) regardless of causality, or deaths during the study including 30 days after treatment discontinuation. A summary of SAEs and other non-serious AEs is located in the Reported Adverse Events section of this report.
Time Frame: Baseline through study completion up to 6 cycles (21-day cycle each) and 30-day safety follow-up
Population: Randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Enzastaurin/Pemetrexed/Carboplatin | Pemetrexed/Carboplatin | Docetaxel/Carboplatin
Number analyzed (Participants) | 67 | 72 | 70
Participants
  AEs | 63 | 70 | 69
  SAEs | 35 | 20 | 26
  Deaths Due to AEs | 3 | 5 | 4

5. Secondary Outcome: Change From Baseline in Total Functional Assessment of Cancer Therapy-Lung (FACT-L) Scale
Description: The FACT-L version 4 scale is used to assess health-related quality of life (HRQoL) in participants with lung cancer. The FACT-L has 5 subscales: Physical Well-Being (PWB), Social and Family Well-Being (SFWB) and Functional Well-Being (FWB) subscales which include 7 items each, Emotional Well-Being (EWB) subscale which includes 6 items, and a Lung-Cancer Specific (LCS) subscale which include 7 items. Total FACT-L is the sum of all 5 subscales. Each item is scored from 0 to 4 giving a total overall score from 0 equal to "worst quality of life" to 136 equal to "best quality of life". The Least Square (LS) mean was calculated using an analysis of covariance (ANCOVA) model adjusted for change scores and baseline scores.
Time Frame: Baseline, Cycle 1 (Week 3), Cycle 2 (Week 6), Cycle 3 (Week 9), Cycle 4 (Week 12), Cycle 5 (Week 15) and Cycle 6 (Week 18) [21-day cycle each]
Population: Randomized participants with non-missing FACT-L data both at baseline and at the specified cycle.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Enzastaurin/Pemetrexed/Carboplatin | Pemetrexed/Carboplatin | Docetaxel/Carboplatin
Number analyzed (Participants) | 45 | 50 | 42
units on a scale
  Cycle 1 (Week 3): number analyzed (Participants) | 43 | 47 | 42
  Cycle 1 (Week 3) | -3.98 (1.86) | 1.12 (1.78) | -3.33 (1.88)
  Cycle 2 (Week 6): number analyzed (Participants) | 45 | 50 | 37
  Cycle 2 (Week 6) | -3.25 (2.19) | -1.54 (2.08) | -2.16 (2.42)
  Cycle 3 (Week 9): number analyzed (Participants) | 35 | 37 | 30
  Cycle 3 (Week 9) | 0.39 (2.30) | 0.64 (2.25) | -1.93 (2.49)
  Cycle 4 (Week 12): number analyzed (Participants) | 32 | 39 | 31
  Cycle 4 (Week 12) | 0.31 (2.47) | 3.54 (2.23) | -0.81 (2.50)
  Cycle 5 (Week 15): number analyzed (Participants) | 25 | 33 | 28
  Cycle 5 (Week 15) | 1.89 (2.95) | -0.26 (2.57) | -4.69 (2.79)
  Cycle 6 (Week 18): number analyzed (Participants) | 16 | 25 | 16
  Cycle 6 (Week 18) | 7.38 (3.54) | -0.83 (2.84) | 3.38 (3.54)
Statistical Analysis 1: Comparison: Enzastaurin/Pemetrexed/Carboplatin vs Docetaxel/Carboplatin; Test type: Superiority or Other; p = 0.96, ANCOVA — P-value is for the change in Total FACT-L at Cycle 1 (Week 3)
Statistical Analysis 2: Comparison: Pemetrexed/Carboplatin vs Docetaxel/Carboplatin; Test type: Superiority or Other; p = 0.15, ANCOVA — P-value is for the change in Total FACT-L at Cycle 1 (Week 3)
Statistical Analysis 3: Comparison: Enzastaurin/Pemetrexed/Carboplatin vs Docetaxel/Carboplatin; Test type: Superiority or Other; p = 0.92, ANCOVA — P-value is for the change in Total FACT-L at Cycle 2 (Week 6)
Statistical Analysis 4: Comparison: Pemetrexed/Carboplatin vs Docetaxel/Carboplatin; Test type: Superiority or Other; p = 0.97, ANCOVA — P-value is for the change in Total FACT-L at Cycle 2 (Week 6)
Statistical Analysis 5: Comparison: Enzastaurin/Pemetrexed/Carboplatin vs Docetaxel/Carboplatin; Test type: Superiority or Other; p = 0.71, ANCOVA — P-value is for the change in Total FACT-L at Cycle 3 (Week 9)
Statistical Analysis 6: Comparison: Pemetrexed/Carboplatin vs Docetaxel/Carboplatin; Test type: Superiority or Other; p = 0.66, ANCOVA — P-value is for the change in Total FACT-L at Cycle 3 (Week 9)
Statistical Analysis 7: Comparison: Enzastaurin/Pemetrexed/Carboplatin vs Docetaxel/Carboplatin; Test type: Superiority or Other; p = 0.93, ANCOVA — P-value is for the change in Total FACT-L at Cycle 4 (Week 12)
Statistical Analysis 8: Comparison: Pemetrexed/Carboplatin vs Docetaxel/Carboplatin; Test type: Superiority or Other; p = 0.33, ANCOVA — P-value is for the change in Total FACT-L at Cycle 4 (Week 12)
Statistical Analysis 9: Comparison: Enzastaurin/Pemetrexed/Carboplatin vs Docetaxel/Carboplatin; Test type: Superiority or Other; p = 0.19, ANCOVA — P-value is for the change in Total FACT-L at Cycle 5 (Week 15)
Statistical Analysis 10: Comparison: Pemetrexed/Carboplatin vs Docetaxel/Carboplatin; Test type: Superiority or Other; p = 0.40, ANCOVA — P-value is for the change in Total FACT-L at Cycle 5 (Week 15)
Statistical Analysis 11: Comparison: Enzastaurin/Pemetrexed/Carboplatin vs Docetaxel/Carboplatin; Test type: Superiority or Other; p = 0.63, ANCOVA — P-value is for the change in Total FACT-L at Cycle 6 (Week 18)
Statistical Analysis 12: Comparison: Pemetrexed/Carboplatin vs Docetaxel/Carboplatin; Test type: Superiority or Other; p = 0.55, ANCOVA — P-value is for the change in Total FACT-L at Cycle 6 (Week 18)

6. Secondary Outcome: Change From Baseline in Total Functional Assessment of Cancer Therapy -Taxane (FACT-Taxane) Scale
Description: The FACT-Taxane version 4 scale is used to assess HRQoL in participants receiving taxane chemotherapy. The FACT-taxane has 5 subscales: PWB, SFWB, and FWB subscales which include 7 items each, EWB subscale which includes 6 items, and a taxane subscale which include 16 items and has two domains (neurotoxicity and taxane). Total FACT-Taxane is the sum of all the 5 subscales. Each item is scored from 0 to 4 giving a total overall score from 0 "worst quality of life" to 172 "best quality of life". The LS mean was calculated using an ANCOVA model adjusted for change scores and baseline scores.
Time Frame: as for outcome 5
Population: Randomized participants with non-missing FACT-Taxane data both at baseline and at the specified cycle.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Enzastaurin/Pemetrexed/Carboplatin | Pemetrexed/Carboplatin | Docetaxel/Carboplatin
Number analyzed (Participants) | 45 | 50 | 43
units on a scale
  Cycle 1 (Week 3): number analyzed (Participants) | 43 | 48 | 43
  Cycle 1 (Week 3) | -3.16 (2.20) | -0.78 (2.08) | -2.17 (2.20)
  Cycle 2 (Week 6): number analyzed (Participants) | 45 | 50 | 38
  Cycle 2 (Week 6) | -6.22 (2.90) | -5.66 (2.76) | -3.13 (3.16)
  Cycle 3 (Week 9): number analyzed (Participants) | 35 | 36 | 30
  Cycle 3 (Week 9) | -1.89 (3.35) | -1.52 (3.32) | -4.40 (3.62)
  Cycle 4 (Week 12): number analyzed (Participants) | 32 | 39 | 30
  Cycle 4 (Week 12) | -2.28 (3.65) | -0.77 (3.29) | -2.58 (3.74)
  Cycle 5 (Week 15): number analyzed (Participants) | 25 | 33 | 28
  Cycle 5 (Week 15) | -2.52 (3.71) | -3.11 (3.24) | -7.74 (3.51)
  Cycle 6 (Week 18): number analyzed (Participants) | 17 | 25 | 16
  Cycle 6 (Week 18) | 2.77 (3.93) | -2.81 (3.26) | -0.34 (4.06)
Statistical Analysis 1: Comparison: Enzastaurin/Pemetrexed/Carboplatin vs Docetaxel/Carboplatin; Test type: Superiority or Other; p = 0.93, ANCOVA — P-value is for the change in Total FACT-Taxane at Cycle 1 (Week 3)
Statistical Analysis 2: Comparison: Pemetrexed/Carboplatin vs Docetaxel/Carboplatin; Test type: Superiority or Other; p = 0.86, ANCOVA — P-value is for the change in Total FACT-Taxane at Cycle 1 (Week 3)
Statistical Analysis 3: Comparison: Enzastaurin/Pemetrexed/Carboplatin vs Docetaxel/Carboplatin; Test type: Superiority or Other; p = 0.69, ANCOVA — P-value is for the change in Total FACT-Taxane at Cycle 2 (Week 6)
Statistical Analysis 4: Comparison: Pemetrexed/Carboplatin vs Docetaxel/Carboplatin; Test type: Superiority or Other; p = 0.77, ANCOVA — P-value is for the change in Total FACT-Taxane at Cycle 2 (Week 6)
Statistical Analysis 5: Comparison: Enzastaurin/Pemetrexed/Carboplatin vs Docetaxel/Carboplatin; Test type: Superiority or Other; p = 0.83, ANCOVA — P-value is for the change in Total FACT-Taxane at Cycle 3 (Week 9)
Statistical Analysis 6: Comparison: Pemetrexed/Carboplatin vs Docetaxel/Carboplatin; Test type: Superiority or Other; p = 0.78, ANCOVA — P-value is for the change in Total FACT-Taxane at Cycle 3 (Week 9)
Statistical Analysis 7: Comparison: Enzastaurin/Pemetrexed/Carboplatin vs Docetaxel/Carboplatin; Test type: Superiority or Other; p = 1.00, ANCOVA — P-value is for the change in Total FACT-Taxane at Cycle 4 (Week 12)
Statistical Analysis 8: Comparison: Pemetrexed/Carboplatin vs Docetaxel/Carboplatin; Test type: Superiority or Other; p = 0.91, ANCOVA — P-value is for the change in Total FACT-Taxane at Cycle 4 (Week 12)
Statistical Analysis 9: Comparison: Enzastaurin/Pemetrexed/Carboplatin vs Docetaxel/Carboplatin; Test type: Superiority or Other; p = 0.49, ANCOVA — P-value is for the change in Total FACT-Taxane at Cycle 5 (Week 15)
Statistical Analysis 10: Comparison: Pemetrexed/Carboplatin vs Docetaxel/Carboplatin; Test type: Superiority or Other; p = 0.53, ANCOVA — P-value is for the change in Total FACT-Taxane at Cycle 5 (Week 15)
Statistical Analysis 11: Comparison: Enzastaurin/Pemetrexed/Carboplatin vs Docetaxel/Carboplatin; Test type: Superiority or Other; p = 0.80, ANCOVA — P-value is for the change in Total FACT-Taxane at Cycle 6 (Week 18)
Statistical Analysis 12: Comparison: Pemetrexed/Carboplatin vs Docetaxel/Carboplatin; Test type: Superiority or Other; p = 0.85, ANCOVA — P-value is for the change in Total FACT-Taxane at Cycle 6 (Week 18)

7. Secondary Outcome: Overall Survival (OS)
Description: OS was the duration from the date of randomization to the date of death from any cause. For participants who were alive, OS was censored at the date of last follow-up visit or at the date of last contact.
Time Frame: Baseline to date of death from any cause up to 35 months
Population: All randomized participants. Sixteen (16) participants in Enzastaurin/Pemetrexed/Carboplatin group, 20 participants in Pemetrexed/Carboplatin group, and 19 participants in Docetaxel/Carboplatin group were censored for analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enzastaurin/Pemetrexed/Carboplatin | Pemetrexed/Carboplatin | Docetaxel/Carboplatin
Number analyzed (Participants) | 56 | 54 | 53
months | 7.2 [5.7 to 11.2] | 12.7 [9.3 to 17.0] | 9.2 [5.9 to 10.7]
Statistical Analysis 1: Comparison: Enzastaurin/Pemetrexed/Carboplatin vs Docetaxel/Carboplatin; Test type: Superiority or Other; p = 0.87, Log Rank
Statistical Analysis 2: Comparison: Pemetrexed/Carboplatin vs Docetaxel/Carboplatin; Test type: Superiority or Other; p = 0.05, Log Rank

8. Secondary Outcome: Number of Participants With Complete Response (CR) or Partial Response (PR) [Tumor Response]
Description: Response was defined using RECIST, version 1.0 criteria. Participants with a best response of CR or PR were considered to have had a tumor response. CR was defined as the disappearance of all target lesions. PR was defined as having at least a 30% decrease in sum of longest diameter of target lesions.
Time Frame: Baseline to measured PD up to 22.3 months
Population: All randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Enzastaurin/Pemetrexed/Carboplatin | Pemetrexed/Carboplatin | Docetaxel/Carboplatin
Number analyzed (Participants) | 72 | 74 | 72
Participants | 9 | 16 | 19

9. Secondary Outcome: Duration of CR or PR (Duration of Response)
Description: The duration of a CR or PR was defined as the time from first objective status assessment of CR or PR to the first time of progression or death due to any cause. Response was defined using RECIST, version 1.0 criteria. CR was defined as the disappearance of all target lesions. PR was defined as having at least a 30% decrease in sum of longest diameter of target lesions.
Time Frame: Date of first response to the date of progression or death due to any cause up to 22.3 months
Population: All randomized participants. 63 participants in Enzastaurin/Pemetrexed/Carboplatin group, 58 participants in Pemetrexed/Carboplatin group, and 53 participants in Docetaxel/Carboplatin group were censored for analysis.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Enzastaurin/Pemetrexed/Carboplatin: Enzastaurin loading dose of 1125 mg or 1200 mg on Day -7 (pre-chemotherapy) followed by 500 mg administered once daily starting from Day -6 until disease progression.
  Pemetrexed 500 mg/m^2 and carboplatin AUC 6 mg*min/mL as an intravenous infusion on Day 1 every 21 days for a maximum of 6 cycles (21-day cycle) or disease progression whichever came first.
Arm/Group | Enzastaurin/Pemetrexed/Carboplatin | Pemetrexed/Carboplatin | Docetaxel/Carboplatin
Number analyzed (Participants) | 9 | 16 | 19
months | 7.4 [3.7 to 8.8] | 9.3 [5.7 to 14.8] | 5.8 [3.3 to 11.3]

10. Secondary Outcome: Time-to-Treatment Failure (TTF)
Description: TTF was defined as the time from randomization to the first observation of PD, death due to any cause, or early discontinuation of treatment. Response was defined using RECIST, version 1.0 criteria. PD was defined as having at least a 20% increase in sum of longest diameter of target lesions. TTF was censored at the date of the last follow-up visit for participants who did not discontinue early, who were still alive, and who have not progressed.
Time Frame: Baseline to stopping treatment up to 14.1 months
Population: All randomized participants. Thirty four (34) participants in Pemetrexed/Carboplatin group and 23 participants in Docetaxel/Carboplatin group were censored for analysis. No participants were censored in Enzastaurin/Pemetrexed/Carboplatin group.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enzastaurin/Pemetrexed/Carboplatin | Pemetrexed/Carboplatin | Docetaxel/Carboplatin
Number analyzed (Participants) | 38 | 51 | 72
months | 2.6 [1.7 to 3.7] | 3.8 [2.8 to 5.1] | 2.6 [1.3 to 3.7]
Statistical Analysis 1: Comparison: Enzastaurin/Pemetrexed/Carboplatin vs Docetaxel/Carboplatin; Test type: Superiority or Other; p = 0.71, Log Rank
Statistical Analysis 2: Comparison: Pemetrexed/Carboplatin vs Docetaxel/Carboplatin; Test type: Superiority or Other; p = 0.04, Log Rank

ADVERSE EVENTS:
Description: Study-specific clinical outcomes due to PD were not considered to be a SAE unless the investigator deemed it related to the use of the study drug.
Arm/Group | Enzastaurin/Pemetrexed/Carboplatin | Pemetrexed/Carboplatin | Docetaxel/Carboplatin
Serious Adverse Events (participants affected / at risk) | 35/67 | 20/72 | 26/70
Other Adverse Events (participants affected / at risk) | 63/67 | 70/72 | 69/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enzastaurin/Pemetrexed/Carboplatin (N=67) | Pemetrexed/Carboplatin (N=72) | Docetaxel/Carboplatin (N=70)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 6 (8)
Arrhythmia (Cardiac disorders) | 3 (3) | 1 (2) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Caecitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 3 (3)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (2) | 1 (1) | 1 (1)
Chest pain (General disorders) | 3 (3) | 0 (0) | 0 (0)
Disease progression (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1)
Localised oedema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Oedema due to cardiac disease (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 1 (1)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 7 (8) | 3 (3) | 2 (3)
Sepsis (Infections and infestations) | 2 (2) | 0 (0) | 4 (4)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 1 (1)
Aspartate aminotransferase (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood calcium decreased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Blood creatinine (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood potassium decreased (Investigations) | 3 (3) | 0 (0) | 0 (0)
Blood sodium decreased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Haemoglobin (Investigations) | 4 (4) | 3 (3) | 2 (2)
Neutrophil count (Investigations) | 1 (1) | 0 (0) | 3 (3)
Platelet count (Investigations) | 1 (1) | 0 (0) | 0 (0)
White blood cell count (Investigations) | 3 (3) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 4 (4) | 1 (1) | 5 (5)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 5 (6) | 0 (0) | 3 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Gastric cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 3 (3) | 1 (1)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 3 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 3 (3)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Aortic thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Enzastaurin/Pemetrexed/Carboplatin (N=67) | Pemetrexed/Carboplatin (N=72) | Docetaxel/Carboplatin (N=70)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 4 (15) | 4 (8)
Arrhythmia (Cardiac disorders) | 3 (4) | 4 (4) | 4 (4)
Dry eye (Eye disorders) | 4 (4) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 4 (6) | 3 (3) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 9 (9) | 5 (6) | 6 (8)
Constipation (Gastrointestinal disorders) | 17 (22) | 25 (26) | 17 (19)
Diarrhoea (Gastrointestinal disorders) | 18 (29) | 10 (12) | 19 (23)
Dyspepsia (Gastrointestinal disorders) | 6 (6) | 2 (2) | 7 (7)
Nausea (Gastrointestinal disorders) | 34 (57) | 32 (52) | 24 (40)
Stomatitis (Gastrointestinal disorders) | 6 (6) | 14 (16) | 13 (15)
Vomiting (Gastrointestinal disorders) | 16 (23) | 18 (20) | 15 (19)
Chest pain (General disorders) | 9 (12) | 13 (15) | 8 (8)
Fatigue (General disorders) | 28 (46) | 39 (55) | 35 (63)
Localised oedema (General disorders) | 2 (5) | 5 (5) | 2 (2)
Oedema peripheral (General disorders) | 9 (10) | 14 (16) | 7 (8)
Pyrexia (General disorders) | 5 (5) | 8 (8) | 7 (8)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 6 (10)
Rhinitis (Infections and infestations) | 2 (4) | 7 (10) | 3 (3)
Vaginal infection (Infections and infestations) | 2/28 (3) | 1/32 (1) | 0/29 (0)
Alanine aminotransferase (Investigations) | 3 (4) | 9 (10) | 1 (1)
Aspartate aminotransferase (Investigations) | 3 (4) | 4 (7) | 2 (2)
Blood albumin decreased (Investigations) | 2 (2) | 6 (10) | 6 (7)
Blood alkaline phosphatase (Investigations) | 3 (3) | 2 (2) | 4 (11)
Blood creatinine (Investigations) | 2 (2) | 7 (9) | 4 (4)
Blood magnesium decreased (Investigations) | 2 (3) | 7 (8) | 3 (3)
Blood potassium decreased (Investigations) | 6 (9) | 8 (10) | 6 (8)
Blood potassium increased (Investigations) | 2 (2) | 4 (5) | 3 (3)
Blood sodium decreased (Investigations) | 6 (6) | 6 (7) | 4 (6)
Haemoglobin (Investigations) | 40 (99) | 53 (132) | 34 (59)
Neutrophil count (Investigations) | 33 (88) | 37 (114) | 46 (138)
Platelet count (Investigations) | 37 (116) | 43 (151) | 18 (41)
Weight decreased (Investigations) | 7 (7) | 5 (5) | 2 (2)
White blood cell count (Investigations) | 23 (63) | 29 (99) | 21 (65)
Decreased appetite (Metabolism and nutrition disorders) | 12 (16) | 12 (13) | 19 (27)
Dehydration (Metabolism and nutrition disorders) | 14 (15) | 6 (6) | 8 (8)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (9) | 13 (32) | 7 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (9) | 5 (8) | 7 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 12 (14) | 6 (7)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 12 (16) | 9 (10) | 10 (11)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 5 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (5) | 7 (7) | 5 (8)
Dizziness (Nervous system disorders) | 12 (14) | 6 (8) | 7 (7)
Dysgeusia (Nervous system disorders) | 6 (7) | 7 (7) | 14 (15)
Headache (Nervous system disorders) | 5 (5) | 5 (5) | 4 (4)
Peripheral sensory neuropathy (Nervous system disorders) | 8 (8) | 9 (10) | 13 (14)
Syncope (Nervous system disorders) | 4 (4) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 4 (4) | 5 (5) | 4 (5)
Depressed mood (Psychiatric disorders) | 2 (2) | 5 (5) | 5 (5)
Insomnia (Psychiatric disorders) | 8 (8) | 8 (8) | 14 (15)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 4 (4) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 0/39 (0) | 2/40 (2) | 1/41 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 17 (19) | 12 (15)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 15 (17) | 16 (19) | 13 (16)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 5 (5) | 3 (3)
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 5 (8) | 5 (6) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (4) | 6 (6) | 20 (22)
Dry skin (Skin and subcutaneous tissue disorders) | 5 (5) | 2 (2) | 3 (3)
Exfoliative rash (Skin and subcutaneous tissue disorders) | 7 (9) | 15 (15) | 5 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 7 (7) | 3 (4)
Hypotension (Vascular disorders) | 7 (7) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days